CLINICAL TRIAL: NCT04777357
Title: A 6-week, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study of the Efficacy and Safety of Cariprazine in Pediatric Subjects (10 to 17 Years of Age) in the Treatment of Depressive Episodes Associated With Bipolar I Disorder
Brief Title: A Study to Assess Change in Disease Activity and Adverse Events (AEs) With Cariprazine in the Treatment of Depressive Episodes in Pediatric Participants Participants (10 to 17 Years of Age) With Bipolar I Disorder.
Acronym: 3112 Ped BPD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3112-301-001; 2020-004758-32 (EudraCT Number)
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Depression; Bipolar I Disorder
Keywords: Depression; RGH-188; Bipolar I Disorder; Vraylar; Cariprazine
MeSH Terms: conditions — Depression | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cariprazine (Experimental): Participants will receive flexible dose Cariprazine over a 6 week treatment period.
  Interventions: Drug: Cariprazine
- Placebo (Placebo Comparator): Participants will receive Placebo over a 6 week treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cariprazine — Oral Capsule
  Other Names: Vraylar
  Arms: Cariprazine
Drug: Placebo — Oral Capsule
  Arms: Placebo

SUMMARY:
Bipolar disorder is a severe chronic mood disorder that affects up to 4% of the adult population and 1.8% of the pediatric population in the United States. The treatment of the depressive episodes of bipolar disorder in the pediatric population has not been as widely studied as the treatment of depressive episodes in bipolar disorder in adults, therefore pharmacotherapeutic options are limited. Given the change in disease state and safety demonstrated in adults with depressive episodes associated with bipolar I disorder, the purpose of this study is to evaluate the change in disease state and safety of cariprazine in the treatment of depressive episodes associated with bipolar I disorder in the pediatric population.

Cariprazine is an approved drug for the treatment of depressive episodes in adult participants with bipolar I disorder. Study doctors put participants in 1 of 2 groups, called treatment arms. There is a 1 in 2 chance that a participant will be assigned to placebo. Around 380 Participants ages 10-17 years with bipolar I disorder will be enrolled in approximately 60 sites worldwide.

Participants receiving the study drug will receive Dose A or B of Cariprazine based on age and weight. At Week 3, participants with insufficient response will have their dose increased to Dose B or Dose C, while participants with sufficient response will continue receiving the Dose A or B for the remainder of the treatment period. The treatment period will be followed by a safety follow-up (SFU) period for 4 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular weekly visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) primary diagnosis of bipolar I disorder as confirmed by Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL).
* Current depressive episode is more than 2 weeks and less than 12 months in duration.
* Participant has a lifetime history of at least one manic episode.
* Children's Depression Rating Scale - Revised (CDRS-R) score > = 45 at Visit 1 and Visit 2.
* Young-Mania Rating Scale (YMRS) score < = 12 with YMRS Item 1 (elevated mood) score < = 2 at Visit 1 and Visit 2.
* Clinical Global Impression-Severity (CGI-S) scale score of > = 4 (moderately ill) at Visit 1 and Visit 2.

Exclusion Criteria:

* Participants with DSM-5 diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, brief psychotic disorder, psychotic disorder due to another medical condition, PTSD, antisocial personality disorder, or borderline personality disorder.
* Participant has a history of meeting DSM-5 diagnosis for any substance-related disorder (except caffeine- and tobacco-related) within the 3 months before Screening Visit 1.
* History of serotonin syndrome or neuroleptic malignant syndrome.
* Four or more episodes of a mood disturbance within the 12 months before Visit 1.
* DSM-5 diagnosis of intellectual disability (IQ < 70), autism spectrum disorders, or documented history of chromosomal disorder with developmental impairment.
* History of seizures, with the exception of febrile seizures.
* Significant head trauma, history of tumor of the CNS, or any other condition that predisposes to seizures.
* Participant requires concomitant treatment with moderate or strong CYP3A4 inhibitors or with any CYP3A4 inducers.
* Participant requires concomitant treatment with any prohibited medication, supplement, or herbal product, including any psychotropic drug or any drug with psychotropic activity or with a potentially psychotropic component.
* Use of a depot antipsychotic within 2 cycles of their respective dosing interval prior to Screening Visit 1.
* Treatment with clozapine in a dose of >= 50 mg/d in the past 2 years.
* History of or any current ocular disease including, but not limited to, retinal detachment, intraocular surgery, laser treatment, glaucoma, cataracts, or clinically significant ocular trauma (with the exception of refractive errors).

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 380 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Baseline (Week 0) to Week 10
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a casual relationship with this treatment. The investigator assesses the relationship of each event to the use of the study. A serious adverse event (SAE) is an event that results in death, is life threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event, that based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/ treatment emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of the study drug.
Abnormal Change from Baseline in Vital Signs | Baseline (Week 0) to Week 10
  Change in vital signs like systolic and diastolic blood pressure will be assessed.
Number of Participants with Incidence of Abnormal Clinical Laboratory Test Results | Baseline (Week 0) to Week 6
  Number of participants with incidence of abnormal clinical laboratory test results like hematology will be assessed.
Change in Electrocardiogram (ECG) | Baseline (Week 0) to Week 6
  12 -lead resting ECGs will be recorded. Parameters include RR interval, PR interval, QT interval, and QRS duration.
Change From Baseline in Simpson-Angus Scale (SAS) | Baseline (Week 0) to Week 6
  SAS is a 10-item rating scale for assessment of antipsychotic-induced parkinsonism in both clinical practice and research settings. Each item ranges from 0 (normal) to 4 (extreme symptoms). The scale consists of 1 item measuring gait (hypokinesia), 6 items measuring rigidity, and 3 items measuring glabella tap, tremor, and salivation, respectively.
Change from Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline (Week 0) to Week 10
  The C-SSRS is a clinician-rated instrument that reports the severity of both suicidal ideation and behavior, with a higher score denoting more severe suicidal ideation and behavior.
Change From Baseline in Barnes Akathisia Rating Scale (BARS) | Baseline (Week 0) to Week 6
  BARS is a 4-item rating scale used to assess drug-induced akathisia. The scale comprises items for rating the observable restless movements that characterize the condition, the subjective awareness of restlessness, and any distress associated with the akathisia (each on a 4-point scale from normal [0] to severe [3]). In addition, there is a global severity for akathisia rated on a 6-point scale (absent [0] to severe akathisia [5]).
Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) | Baseline (Week 0) to Week 6
  AIMS assesses abnormal involuntary movements, such as tardive dyskinesia, associated with antipsychotic drugs; it measures facial, oral, extremities, and trunk movements, as well as the participant's awareness of abnormal movements. The first 10 items are rated on a none (0) to severe (4) scale. There are an additional 2 items on dental status that are answered yes or no.
Change in Children's Depression Rating Scale - Revised (CDRS-R) Total Score | Baseline (Week 0) to Week 6
  The CDRS-R is a 17-item clinician-administered scale specifically developed for the assessment of depressive symptoms in children and adolescents. Total scores range from 17 to 113. In general, scores below 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, and scores of 40 to 60 indicate moderate depression. The CDRS-R will be administered by a clinician with extensive professional training in mental illness.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (77):
- United States (65):
  - Pillar Clinical Research /ID# 226504, Bentonville, Arkansas
  - Advanced Research Center /ID# 227073, Anaheim, California
  - Care Access Research /ID# 226316, Beverly Hills, California
  - ProScience Research Group /ID# 226223, Culver City, California
  - National Institute of Clinical Research - Garden Grove /ID# 262835, Garden Grove, California
  - Duplicate_Alliance for Research - Long Beach /ID# 226522, Long Beach, California
  - CHOC Children's Hospital /ID# 260298, Orange, California
  - ATP Clinical Research- Orange /ID# 253719, Orange, California
  - Prospective Research Innovations Inc /ID# 240774, Rancho Cucamonga, California
  - Inland Psychiatric Medical Group /ID# 274621, Redlands, California
  - University of California Davis Health /ID# 268306, Sacramento, California
  - University of California, San Diego Department of Psychiatry /ID# 226463, San Diego, California
  - Lumos Clinical Research Center /ID# 262805, San Jose, California
  - Pacific Clinical Research Management Group /ID# 227075, Upland, California
  - D&H Doral Research Center-Doral /ID# 255458, Doral, Florida
  - Advanced Research Institute of Miami /ID# 228222, Homestead, Florida
  - Columbus Clinical Services, Llc /Id# 229792, Miami, Florida
  - G+C Research Group, LLC /ID# 261399, Miami, Florida
  - Florida Research Center, Inc. /ID# 240775, Miami, Florida
  - South Florida Research Ph I-IV /ID# 240778, Miami Springs, Florida
  - Medical Research Group of Central Florida /ID# 256757, Orange City, Florida
  - APG Research, LLC /ID# 226519, Orlando, Florida
  - Nova Psychiatry Inc. /ID# 270892, Orlando, Florida
  - Panhandle Research and Medical Clinic, LLC /ID# 268522, Pensacola, Florida
  - D&H Tamarac Research Center /ID# 250434, Tamarac, Florida
  - University of South Florida- Neuroscience Institute /ID# 246508, Tampa, Florida
  - Atlanta Center for Medical Research /ID# 226480, Atlanta, Georgia
  - CenExcel iResearch LLC /ID# 228695, Decatur, Georgia
  - Atlanta Behavioral Research, LLC /ID# 226486, Dunwoody, Georgia
  - Sleep Care Research Institute d/b/a Clinical Research Institute /ID# 226371, Stockbridge, Georgia
  - Denali Health Atlanta, LLC /ID# 278167, Stone Mountain, Georgia
  - Duplicate_Ascension St. Elizabeth /ID# 240772, Chicago, Illinois
  - Baber Research Group /ID# 232279, Naperville, Illinois
  - Advanced Quality Medical Research /ID# 272902, Orland Park, Illinois
  - Indiana University /ID# 260705, Indianapolis, Indiana
  - Benchmark Research /ID# 260714, Shreveport, Louisiana
  - The Kennedy Krieger Institute /ID# 226509, Baltimore, Maryland
  - Med Clinical Research Partners LLC /ID# 240773, Irvington, New Jersey
  - Duplicate_NeuroCognitive and Behavioral Institute, Inc /ID# 227077, Mount Arlington, New Jersey
  - UB Department of Psychiatry /ID# 226373, Buffalo, New York
  - New Dawn Psychiatric Services PLLC /ID# 229782, Kinston, North Carolina
  - Quest Therapeutics of Avon Lake /ID# 226349, Avon Lake, Ohio
  - University of Cincinnati /ID# 226465, Cincinnati, Ohio
  - CincyScience /ID# 226318, West Chester, Ohio
  - IPS Research Company /ID# 227072, Oklahoma City, Oklahoma
  - SP Research, PLLC /ID# 259428, Oklahoma City, Oklahoma
  - Cutting Edge Research Group /ID# 240777, Oklahoma City, Oklahoma
  - Paradigm Research Professionals /ID# 260719, Oklahoma City, Oklahoma
  - Sooner Clinical Research /ID# 226384, Oklahoma City, Oklahoma
  - BioBehavioral Research of Austin /ID# 227076, Austin, Texas
  - Beaumont Psychiatric Clinic /ID# 267484, Beaumont, Texas
  - Houston Clinical Trials - Bellaire /ID# 274189, Bellaire, Texas
  - Texas Research Group /ID# 270050, Coppell, Texas
  - Relaro Medical Trials /ID# 227156, Dallas, Texas
  - Earle Research /ID# 253782, Friendswood, Texas
  - McGovern Medical School /ID# 240779, Houston, Texas
  - Southwest Biomed Research Center LLC /ID# 226340, Houston, Texas
  - Kaleidoscope Clinical Research /ID# 277650, Houston, Texas
  - Red Oak Psychiatry Associates /ID# 240776, Houston, Texas
  - Livingspring Family Medical Center /ID# 262706, Mansfield, Texas
  - AIM Trials /ID# 226367, Plano, Texas
  - Perceptive Pharma Research /ID# 262219, Richmond, Texas
  - Family Psychiatry of The Woodlands /ID# 226290, The Woodlands, Texas
  - Pantheon Clinical Research /ID# 270879, Bountiful, Utah
  - Core Clinical Research /ID# 226374, Everett, Washington
- Puerto Rico (2):
  - Dr. Samuel Sanchez PSC /ID# 245952, Caguas
  - GCM Medical Group PSC /ID# 245951, San Juan
- Russia (10):
  - Clinica of Glazunova /ID# 229416, Krasnodar, Krasnodarskiy Kray
  - Duplicate_Scientific Centre of Personalized Medicine /ID# 226380, Moscow, Moscow
  - Duplicate_Central Clinical Psychiatric Hospital /ID# 226381, Moscow, Moscow
  - Orenburg Regional Clinical Psychiatric Hospital #1 /ID# 226462, Orenburg, Orenburg Oblast
  - Psychotherapeutics Center Podderzhka /ID# 226348, Stavropol, Stavropol Kray
  - Clinical Psychiatry Hospital #1 of Nizhniy Novgorod /ID# 226226, Nizhny Novgorod
  - Psychiatric hospital #1 /ID# 226516, Saint Petersburg
  - National Medical Research Center of Psychiatry and Neurology n.a. V.M. Bekhterev /ID# 226515, Saint Petersburg
  - Medgard Clinic /ID# 228598, Saratov
  - Saratov City Clinical Hospital #2 n.a. V. I. Razumovsky /ID# 226222, Saratov

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=3112-301-001